CLINICAL TRIAL: NCT02476045
Title: First-line FOLFOX-4 Plus Panitumumab Followed by 5-FU/LV Plus Panitumumab or Single-agent Panitumumab as Maintenance Therapy in Patients With RAS Wild-type, Metastatic Colorectal Cancer: the VALENTINO Study
Brief Title: Panitumumab-based Maintenance in Patients With RAS Wild-type, Metastatic Colorectal Cancer (Valentino)
Acronym: Valentino
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT 70/15
Record Dates: First submitted 2015-06-11; First posted 2015-06-19 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; RAS wild-type; maintenance therapy; panitumumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Panitumumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Active Comparator): Induction phase with panitumumab as 1 hour intravenous infusion at the dosage of 6 mg/kg, given every two weeks, plus FOLFOX-4 chemotherapy as standard guidelines.
  Maintenance therapy with 5-FU/LV (De Gramont regimen) plus panitumumab given at 6 mg/Kg every two weeks until progressive disease, unacceptable toxicity or informed consent withdrawal
  Interventions: Drug: 5-fluorouracil,leucovorin,panitumumab; Drug: Oxaliplatin, 5-fluorouracil,leucovorin,panitumumab
- ARM B (Experimental): Induction phase with panitumumab as 1 hour intravenous infusion at the dosage of 6 mg/kg, given every two weeks, plus FOLFOX-4 chemotherapy as standard guidelines.
  Maintenance therapy with panitumumab alone given at 6 mg/Kg every two weeks until progressive disease, unacceptable toxicity or informed consent withdrawal
  Interventions: Drug: panitumumab; Drug: Oxaliplatin, 5-fluorouracil,leucovorin,panitumumab

INTERVENTIONS:
Drug: 5-fluorouracil,leucovorin,panitumumab — Maintenance treatment (ARM A)
  Arms: ARM A
Drug: panitumumab — Maintenance treatment (ARM B)
  Arms: ARM B
Drug: Oxaliplatin, 5-fluorouracil,leucovorin,panitumumab — Induction treatment
  Other Names: FOLFOX-4 + panitumumab

SUMMARY:
Open label, randomized, multicenter, phase II study to compare the efficacy, in terms of non-inferiority of progression-free survival (PFS), of maintenance with panitumumab alone (arm B) as compared to panitumumab with 5-fluorouracil (5-FU) and leucovorin (LV) (arm A) following induction treatment with 5-fluorouracil + leucovorin+oxaliplatin (FOLFOX-4) and panitumumab in patients with RAS wild-type, metastatic colorectal cancer.

The study involves an induction phase with panitumumab as 1 hour intravenous infusion at the dosage of 6 mg/kg, given every two weeks, plus FOLFOX-4 chemotherapy as standard guidelines.

Before start of FOLFOX-4 plus panitumumab, at the time of enrollment, patients will be immediately randomized electronically 1:1 to one of the two maintenance arms. Induction treatment with FOLFOX-4 plus panitumumab will continue until progressive disease, unacceptable toxicity or informed consent withdrawal, or for up to 8 cycles. At the end of induction treatment, in presence of complete or partial response, or stable disease, non-progressing patients will be allocated to one of the two pre-assigned maintenance arms:

A) 5-FU/LV (De Gramont regimen) plus panitumumab given at 6 mg/Kg every two weeks until progressive disease, unacceptable toxicity or informed consent withdrawal B) Panitumumab alone given at 6 mg/Kg every two weeks until progressive disease, unacceptable toxicity or informed consent withdrawal Imaging studies (thorax and abdominal CT or MRI scan) will be performed at baseline (4 weeks prior enrollment) and every 8 weeks (4 cycles) during treatment.

DETAILED DESCRIPTION:
First-line treatment of metastatic colorectal cancer should be administered according to the individual situation, patients' needs, therapeutic preconditions (e.g. neurotoxicity following adjuvant oxaliplatin-based chemotherapy), biomarkers and aggressiveness of the disease.

The OPTIMOX1 trial showed an equivalent duration of disease control for a de-escalation / maintenance / reintroduction strategy compared with a treatment until progression strategy for oxaliplatin-based chemotherapy. Continuation of "lightened" fluoropyrimidine-based chemotherapy and bevacizumab represents a standard of care in the maintenance setting.

Panitumumab with FOLFOX-4 chemotherapy represents a standard of care in the treatment of RAS wild-type metastatic colorectal cancer. The question whether the maintenance strategy might apply also to panitumumab in combination with chemotherapy is unknown at present.

As the continuation of chemotherapy plus panitumumab until disease progression was foreseen in the hallmark "PRIME" trial, the question is whether a de-escalation of treatment intensity will not be inferior with respect to resulting time with tumor control, but allow patients a period with less toxicity and gain of quality of life.

However, no data are available at present regarding the optimal maintenance treatment with anti-epidermal growth factor receptor (EGFR) monoclonal antibodies when used in association with first-line chemotherapy.

This is an open label, randomized, multicenter, phase II study to compare the efficacy, in terms of non-inferiority of progression-free survival (PFS), of maintenance with panitumumab alone (arm B) as compared to panitumumab with 5-FU/LV (arm A) following induction treatment with FOLFOX-4 and panitumumab in patients with RAS wild-type, metastatic colorectal cancer.

Secondary endpoints are:

* Safety (according to Common Terminology Criteria for Adverse Events -CTCAE- v 4.03). All Adverse events will be reported according to National Cancer Institute Criteria. The incidence of adverse events will be summarized according to the primary system-organ class (SOC) and within the category defined in the CTCAE v4.03. The summaries will be overall (severity grades 1-4) and for grade ≥3 events and will also report the actions taken in terms of treatment discontinuation. Similar summaries will be made for serious adverse events. The safety set will be considered.
* Quality of life (patients reported outcomes).
* Response rate (RR), duration of response (DR), time to progression (TTP), time to treatment failure (TTF) and overall survival (OS).
* Exploratory endpoints: Archival tumor tissue samples will be collected at baseline. Samples will be sent at Pathology Department of Fondazione IRCCS Istituto Nazionale dei Tumori for exploratory biomarkers substudy A representative formalin-fixed, paraffin-embedded (FFPE) diagnostic tumor specimen, as a tissue block that must have been reviewed by a pathologist to confirm that it contains adequate tumor tissue. In alternative, fifteen 5-micron unstained slides are allowed. Next-generation sequencing (Ion-Torrent) and in-situ hybridization techniques will be performed to identify potential biomarkers of primary resistance. Since the availability of blood-based biomarkers could be particularly useful for prediction of treatment efficacy or acquired resistance to panitumumab, in this study we will collect blood samples (optional) in individual patients (before treatment, every 8 weeks during treatment and at progression) to analyze circulating tumor DNA by digital Polymerase chain reaction (ddPCR) or next generation (NGS) approaches. Moreover, pharmacogenetic studies to predict panitumumab and chemotherapy toxicity are planned.

Treatment involves an induction phase with panitumumab as 1 hour intravenous infusion at the dosage of 6 mg/kg, given every two weeks, plus FOLFOX-4 chemotherapy as standard guidelines.

Before start of FOLFOX-4 plus panitumumab, at the time of enrollment, patients will be immediately randomized electronically 1:1 to one of the two maintenance arms. Induction treatment with FOLFOX-4 plus panitumumab will continue until progressive disease, unacceptable toxicity or informed consent withdrawal, or for up to 8 cycles. At the end of induction treatment, in presence of complete or partial response, or stable disease, non-progressing patients will be allocated to one of the two pre-assigned maintenance arms:

A) 5-FU/LV (De Gramont regimen) plus panitumumab given at 6 mg/Kg every two weeks until progressive disease, unacceptable toxicity or informed consent withdrawal B) Panitumumab alone given at 6 mg/Kg every two weeks until progressive disease, unacceptable toxicity or informed consent withdrawal Imaging studies (thorax and abdominal CT or MRI scan) will be performed at baseline (4 weeks prior enrollment) and every 8 weeks (4 cycles) during treatment.

The sample size is calculated on the basis of a non-inferiority hypothesis of median PFS with panitumumab alone as compared to 5-fluorouracil/leucovorin and panitumumab, taking into account a median PFS of 10 months observed in the PRIME trial. An overall sample size of 224 subjects (112 in the control group and 112 in the study group) achieves 90% power to detect a probability of 50% in the control group and a maximum difference of 15% in the study group, with a significance level of 0.1. The drop-out rate is 15%. The accrual pattern in the two groups is uniform (allocation 1:1).

The study lasts for 24 months of enrollment and 12 months of follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to performance of any study procedure;
2. Age ≥18 years;
3. ECOG Performance Status 0-1;
4. Life expectancy of at least 12 weeks in the opinion of the Investigator;
5. Histologically or cytologically confirmed adenocarcinoma of the colon or rectum, with RAS wild-type status;
6. Metastatic unresectable colorectal cancer not previously treated with standard chemotherapy for advanced or metastatic disease;
7. Measurable or non-measurable metastatic lesion(s), as defined by RECIST version 1.1;
8. Laboratory requirements:

   * Neutrophils >= 1.5 x 109/L, Platelets >= 100 x 109/L, and Haemoglobin >=10g/dL
   * Total bilirubin <= 1.5 time the upper-normal limits (UNL) of the Institutional normal values; ASAT (SGOT) and/or ALAT (SGPT) <= 2.5 x UNL, or <= 5 x UNL in case of liver metastases; alkaline phosphatase <= 2.5 x UNL, <= 5 x UNL in case of liver metastases, <= 10 x UNL in case of bone metastases; LDH <1500 U/L
   * Creatinine clearance (calculated according to Cockcroft and Gault) > 60 mL/min or serum creatinine <=1.5 x upper limit of normal (UNL);
9. Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating center.
10. Archival tumor tissue is required for exploratory research at enrolment.

Exclusion Criteria:

1. Has a serious illness or medical condition(s) including, but not limited to the following:

   1. Other concurrently active malignancies excluding malignancies that are disease free for more than 5 years or carcinoma-in-situ deemed cured by adequate treatment.
   2. Known brain metastasis or leptomeningeal metastasis.
   3. Active infection (ie, body temperature ≥38°C due to infection).
   4. Ascites, pleural effusion or pericardial fluid requiring drainage in last 4 weeks.
   5. Intestinal obstruction, pulmonary fibrosis or interstitial pneumonitis, renal failure, liver failure, or cerebrovascular disorder.
   6. Uncontrolled diabetes.
   7. Myocardial infarction within the last 12 months, severe/unstable angina, symptomatic congestive heart failure New York Heart Association (NYHA) class III or IV
   8. Gastrointestinal hemorrhage.
   9. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or hepatitis B or C.
   10. Autoimmune disorders or history of organ transplantation that require immunosuppressive therapy.
   11. Psychiatric disease that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results.
2. Patients who had received adjuvant oxaliplatin-based chemotherapy and had recurrence during treatment or within 12 months from its completion are excluded. Patients who had received adjuvant fluoropyrimidine mono-therapy and had recurrence during treatment or within 6 months from its completion are excluded.
3. Disease that is deemed potentially resectable after conversion chemotherapy is excluded. In particular, patients must be deemed unresectable by a multidisciplinary team, even when foreseeing a response to treatment. In case of liver metastases, the concept of resectability must take into account both the aim of oncological radicality (R0 resection) and remanent liver function considerations.
4. Treatment with any of the following within the specified time frame prior to study drug administration:

   1. Major surgery within prior 4 weeks (the surgical incision should be fully healed prior to study drug administration).
   2. Any anticancer therapy or investigational agent within prior 4 weeks
   3. Extended field radiation within prior 4 weeks or limited field radiation within prior 2 weeks.
5. Has unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation). In particular, patients with platinum induced neurotoxicity greater than or equal CTCAE Grade 2 should be excluded.
6. Is a pregnant or lactating female, or is planning to become pregnant during treatment and within 2 months after the end of treatment with panitumumab. Women of child-bearing potential with either positive or no pregnancy test at baseline. Women of child-bearing potential or sexually active men not willing to use contraception during study and for at least 2 months after end of treatment with panitumumab. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 3 years
  in terms of progression free survival (from the enrollment)

SECONDARY OUTCOMES:
Safety in terms of number of participants with adverse events. | 3 years
  in terms of number of participants with adverse events.
Quality of life | 3 years
Response rate | 3 years
duration of response | 3 years
time to progression | 3 years
time to treatment failure | 3 years
overall survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei tumori, Milan, MI, Italy

REFERENCES:
- [Derived] Morano F, Corallo S, Lonardi S, Raimondi A, Cremolini C, Rimassa L, Murialdo R, Zaniboni A, Sartore-Bianchi A, Tomasello G, Racca P, Clavarezza M, Adamo V, Perrone F, Gloghini A, Tamborini E, Busico A, Martinetti A, Palermo F, Loupakis F, Milione M, Fuca G, Di Bartolomeo M, de Braud F, Pietrantonio F. Negative Hyperselection of Patients With RAS and BRAF Wild-Type Metastatic Colorectal Cancer Who Received Panitumumab-Based Maintenance Therapy. J Clin Oncol. 2019 Nov 20;37(33):3099-3110. doi: 10.1200/JCO.19.01254. Epub 2019 Sep 20. PMID 31539295
- [Derived] Pietrantonio F, Morano F, Corallo S, Miceli R, Lonardi S, Raimondi A, Cremolini C, Rimassa L, Bergamo F, Sartore-Bianchi A, Tampellini M, Racca P, Clavarezza M, Berenato R, Caporale M, Antista M, Niger M, Smiroldo V, Murialdo R, Zaniboni A, Adamo V, Tomasello G, Giordano M, Petrelli F, Longarini R, Cinieri S, Falcone A, Zagonel V, Di Bartolomeo M, de Braud F. Maintenance Therapy With Panitumumab Alone vs Panitumumab Plus Fluorouracil-Leucovorin in Patients With RAS Wild-Type Metastatic Colorectal Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2019 Sep 1;5(9):1268-1275. doi: 10.1001/jamaoncol.2019.1467. PMID 31268481